CLINICAL TRIAL: NCT02248285
Title: Implementation of a Molecular Diagnostic for Pediatric Acute Gastroenteritis: The FilmArray GI Panel IMPACT Study
Acronym: IMPACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BioFire Diagnostics, LLC (Industry)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: DX-SDY-019839; R01AI104593 (NIH)
Record Dates: First submitted 2014-09-18; First posted 2014-09-25 (Estimated); Results first posted 2017-12-26 (Actual); Last update posted 2017-12-26 (Actual); Status verified 2017-11

CONDITIONS: Infectious Gastroenteritis
Keywords: multiplex; polymerase chain reaction; PCR; BioFire Diagnostics; Infectious gastroenteritis; Diarrheal disease; Emergency department; rapid diagnostics; FilmArray; FilmArray GI Panel
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): FilmArray™ GI Panel testing will be standard of care and provided at no cost. Additional testing may be ordered at the discretion of the clinician.
  Interventions: Device: FilmArray™ Gastrointestinal (GI) Panel
- Pre-intervention (No Intervention): Testing will be at the discretion of the clinician using standard laboratory tests, and specimens will be collected as appropriate for these methods.

INTERVENTIONS:
Device: FilmArray™ Gastrointestinal (GI) Panel — BioFire Diagnostics, LLC (BioFire) has developed a polymerase chain reaction (PCR), high-resolution melting analysis instrument called the FilmArray™ and an associated reagent pouch that together are capable of simultaneously detecting multiple microorganisms in a single sample. The FilmArray™ Gastrointestinal (GI) Panel pouch contains freeze-dried reagents to perform nucleic acid purification and nested, multiplex PCR for the identification of common bacterial, viral, and parasite microorganisms responsible for infectious gastroenteritis. The test was made available for sale in the US and EU following FDA clearance and CE marking in May, 2014
  Arms: Intervention

SUMMARY:
BioFire Diagnostics, LLC (BioFire) has developed the FilmArray Gastrointestinal (GI) Panel, a rapid, easy to use PCR-based in vitro diagnostic test for the identification of 22 common microorganisms responsible for infectious gastroenteritis (http://filmarray.com/the-panels/) from a stool specimen collected in Cary Blair enteric transport media. The test was made available for sale in the US and EU following FDA clearance and CE marking in May, 2014.

The FilmArray GI Panel offers improvements over conventional laboratory testing which include: reduced turnaround time from specimen to result, reduced laboratory labor costs, increased sensitivity and specificity relative to current clinical reference methods, and larger breadth of organism identification than is available using standard methods. Because of these attributes, the results from this test have the potential to enable clinicians to more accurately diagnose and treat GI illness in a reduced time frame.

Collaborators at the University of Utah, Brown University/Lifespan, and BioFire Diagnostics have designed a study to evaluate health outcomes of pediatric subjects presenting to emergency departments with GI illness before and after establishing the FilmArray GI Panel as the standard of care method for stool pathogen analysis. It is hypothesized that the rapid (~ 1 hour turnaround time), sensitive, specific, and comprehensive results provided by the FilmArray GI Panel will allow clinicians to more rapidly diagnose GI illness, initiate appropriate therapy and provide guidance when compared to the pre-implementation period.

ELIGIBILITY:
Inclusion Criteria:

* Children (<18 years) presenting to the ED or onsite urgent care center with symptoms of gastroenteritis (e.g. diarrhea, vomiting, nausea, etc.)
* Duration of symptoms at least 24 hours but < 14 days
* Able to provide stool specimen at time of enrollment or within the next two calendar days
* Parent or guardian able to provide permission and subject able to provide assent, if appropriate

Exclusion Criteria:

* Undefined onset of illness or symptoms for ≥14 days
* Unable to complete questionnaire or give informed consent because of language barrier
* Those unable to provide stool specimen at time of enrollment or within two calendar days
* Previous enrollment in this study

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1545 (Actual)
Dates: Start 2015-04; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Children's Hospital of Los Angeles, Los Angeles, California
  - Children's Mercy Hospital, Kansas City, Missouri
  - Nationwide Children's Hospital, Columbus, Ohio
  - Brown University, Lifespan, Providence, Rhode Island
  - University of Utah, Primary Children's Hospital, Salt Lake City, Utah

REFERENCES:
- [Background] Poritz MA, Blaschke AJ, Byington CL, Allen L, Nilsson K, Jones DE, Thatcher SA, Robbins T, Lingenfelter B, Amiott E, Herbener A, Daly J, Dobrowolski SF, Teng DH, Ririe KM. FilmArray, an automated nested multiplex PCR system for multi-pathogen detection: development and application to respiratory tract infection. PLoS One. 2011;6(10):e26047. doi: 10.1371/journal.pone.0026047. Epub 2011 Oct 19. PMID 22039434
- [Background] FDA. FDA clearance for FilmArray Gastrointestinal Panel, May 2, 2014. http://www.accessdata.fda.gov/cdrh_docs/reviews/K140407.pdf (2014).
- [Derived] Pavia AT, Cohen DM, Leber AL, Daly JA, Jackson JT, Selvarangan R, Kanwar N, Bender JM, Dien Bard J, Festekjian A, Duffy S, Larsen C, Holmberg KM, Bardsley T, Haaland B, Bourzac KM, Stockmann C, Chapin KC, Leung DT. Clinical Impact of Multiplex Molecular Diagnostic Testing in Children With Acute Gastroenteritis Presenting to an Emergency Department: A Multicenter Prospective Study. Clin Infect Dis. 2024 Mar 20;78(3):573-581. doi: 10.1093/cid/ciad710. PMID 38097379

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention | Pre-intervention
Started | 687 | 858
Completed | 586 | 571
Not Completed | 101 | 287

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Pre-intervention | Total
Number analyzed (Participants) | 586 | 571 | 1157
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 586 | 571 | 1157
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 2.7 [1.2 to 7.8] | 3 [1.2 to 7.0] | 2.8 [1.2 to 7.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 272 | 300 | 572
  Male | 314 | 271 | 585
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 586 | 571 | 1157

OUTCOME MEASURES:

1. Primary Outcome: Analysis of Diarrheal Illness Etiologies Identified in Stool Culture Compared to the FilmArray™ Gastrointestinal (GI) Panel
Description: Describing of etiology of diarrheal illness in the study as identified by each method
Time Frame: Seven to ten days after enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Pre-intervention
Number analyzed (Participants) | 586 | 64
Participants | 434 | 19

ADVERSE EVENTS:
Arm/Group | Intervention | Pre-intervention
All-Cause Mortality (participants affected / at risk) | 0/586 | 0/571
Serious Adverse Events (participants affected / at risk) | 0/586 | 0/571
Other Adverse Events (participants affected / at risk) | 0/586 | 0/571

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No